CLINICAL TRIAL: NCT01437176
Title: Treatment of Intertrochanteric Fracture With New Type of Intramedullary Nail
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peifu Tang (Other)
Responsible Party: Sponsor-Investigator, Peifu Tang, Chief, Professor, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PLAGH OD 12
Record Dates: First submitted 2011-09-01; First posted 2011-09-20 (Estimated); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Intertrochanteric Fracture
Keywords: surgery; fixation; intramedullary nail
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Unstable intertrochanteric fracture fixed with novel nail (Experimental): AO/OTA A2 fracture fixed with novel nail
  Interventions: Device: new type of intramedullary nail
- unstable intertrochanteric fracture fixed with PFNA (Experimental): AO/OTA A2 fracture fixed with PFNA
  Interventions: Device: The intramedullary nail of PFNA

INTERVENTIONS:
Device: new type of intramedullary nail — This is a new fixation treat for intertrochanteric fracture.
  Other Names: WEIGAO ORTHOPAEDIC DEVICE CO.LTD.; ZL201020121021.6
  Arms: Unstable intertrochanteric fracture fixed with novel nail
Device: The intramedullary nail of PFNA — It was used very common in treat with intertrochanteric fracture.
  Other Names: AO Foundation; PFNA(proximal femoral nail antirotation)
  Arms: unstable intertrochanteric fracture fixed with PFNA

SUMMARY:
The purpose of this study is to determine whether this new intramedullary fixation is effective in the treatment of intertrochanteric fracture.

DETAILED DESCRIPTION:
With the progress of aging society, elderly patients with intertrochanteric fractures were occurred more and more. The best recommend treatment is surgical treatment of intramedullary fixation. However, existing methods of intramedullary fixation could not be restored the integrated interior support, and it will occur early hip varus. Meanwhile, the varus deformity will no longer develop if the two ends contact with wach other. This new intramedullary fixation device can overcome the existing shortage of intramedullary fixation devices and supporting the inside of the problem. It can prompting the fracture site to obtain a stronger initial stability, improve fracture healing rate, reduce the incidence of varus and allow patients with early weight-bearing walking.

This new type of intramedullary fixation of intertrochanteric fractures of devices, including a proximal femoral anatomy and adapt to proximal femoral nail, proximal femoral nail through the femoral head and distal femur compression screw locking screw, its main features are:

1. The proximal femoral nail was made from titanium, its proximal part is narrow inside and wide outside structure. It looks like a trapezoidal in cross-section. This device was matched with the anatomy of proximal femur and its mechanical reliability.
2. The tip of compression screw was designed thread. It can come through the intramedullary nail, produce slide and sustained pressure.
3. The femoral support screw was made in cylindrical, had a blunt rounded tip. The tip of the femoral support screw was tabling with the groove of compression screw. This design can support interior mechanical stability. At the same time, the support screw from the femoral head and neck compression screw can slide fine-tuning, so it has a direct offset against varus and femoral neck rotating shift to prevent secondary loss of fracture reduction. The screw in the femoral head also can prevent cutting occurs.
4. This device can be used in minimally invasive approach of percutaneous and implanted in body. Reduce reduction time, fracture interference and help the natural healing of fractures.

ELIGIBILITY:
Inclusion Criteria:

* Adult men or women aged 18 years and older (with no upper age limit).
* Fracture of the intertrochanteric fracture confirmed with either anteroposterior and lateral hip radiographs, computed tomography, or magnetic resonance imaging (MRI).
* Operative treatment of fractures within 14 days of presenting to the emergency room.
* Patient was ambulatory prior to fracture, though they may have used an aid such as a cane or a walker.
* Anticipated medical optimalization for operative fixation of the hip.
* Provision of informed consent by patient or legal guardian.
* No other major trauma.

Exclusion Criteria:

* Patients not suitable for internal fixation (i.e., severe osteoarthritis, rheumatoid arthritis, or pathologic fracture).
* Associated major injuries of the lower extremity (i.e., ipsilateral or contralateral fractures of the foot, ankle, tibia, fibula, knee, or femur; dislocations of the ankle, knee, or hip; or femoral head defects or fracture).
* Retained hardware around the affected hip.
* Infection around the hip (i.e., soft tissue or bone).
* Patients with disorders of bone metabolism except osteoporosis (i.e., Paget's disease, renal osteodystrophy, osteomalacia).
* Moderate or severe cognitively impaired patients (i.e., Six Item Screener with 3 or more errors).
* Patients with Parkinson's disease (or dementia) severe enough to increase the likelihood of falling or severe enough to compromise rehabilitation.
* Likely problems, in the judgment of the investigators, with maintaining follow-up. We will, for example, exclude patients with no fixed address, those who report a plan to move out of town in the next year, or intellectually challenged patients without adequate family support

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-09; Primary Completion 2022-09 (Actual); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Postoperative quality of life score | preoperative, six months and one year postoperative
  SF-36 PCS

SECONDARY OUTCOMES:
rate of fracture healing at three months | three months postoperative
  fracture healing condition was checked by radiological examination.
rate of femoral medialization | one year postoperative
  femoral medialization
collodiaphyseal angle | one year postoperative
  collodiaphyseal angle
weight bearing | perioperation
  time of weight bearing
rate of patient satisfaction with treatment | one year postoperative
  1-year VAS satisfaction
Hip function score | preoperative, six months and one year postoperative
  OHS
time of surgical during | Perioperative
  The time from the beginning to the end of the surgery
fluoroscopy time | intraoperative
  Duration of fluoroscopy
rate of complications related to implant | one year
  cut out, nonunion, implant breakage/failure, infection

CONTACTS AND LOCATIONS:
Overall Officials: Tang Peifu, Study Chair — Chinese PLA General Hospital
Locations (1):
- Orthopedics department; The General Hospital of the People's Liberation Army, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Nie S, Li J, Liu X, Liu J, Wu X, Tang P, Zhao Y, Li M, Zhang L. The clinical efficacy of Medial Sustain Nail(MSN) and Proximal femoral nail anti-rotation(PFNA) for fixation of medial comminuted trochanteric fractures: a prospective randomized controlled trial. Int Orthop. 2024 Aug;48(8):2189-2200. doi: 10.1007/s00264-024-06220-6. Epub 2024 May 21. PMID 38772935